CLINICAL TRIAL: NCT07063108
Title: Efficacy and Safety of S-ketamine Hydrochloride Injection in Elderly Patients Undergoing Elective Non-cardiac Surgery: a Multicenter, Randomized, Placebo Controlled Clinical Trials（ESSENCE）
Brief Title: Efficacy and Safety of S-ketamine in Elderly Patients Undergoing Non-cardiac Surgery: a RCT（ESSENCE）
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director of Anesthesia Department, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-698
Record Dates: First submitted 2024-11-27; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (esketamine injection) (Experimental): Test group (esketamine injection group)： Intravenous infusion of esketamine: after induction, a single dose of 0.25 mg/kg before skin incision，and continuous 0.125 mg/kg/h until 30 min before surgery was stopped.
  Interventions: Drug: Esketamine hydrochloride
- Control group (placebo: saline) (Placebo Comparator): Control group (placebo: saline): after induction, a single intravenous infusion of an equal amount of 0.9% saline before skin incision, followed by a continuous infusion at the same rate as the test group until 30 min before surgery was stopped.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Esketamine hydrochloride — Intravenous infusion of esketamine: after induction, a single dose of 0.25 mg/kg before skin incision，and continuous 0.125 mg/kg/h until 30 min before surgery was stopped.
  Arms: Test group (esketamine injection)
Drug: Saline — after induction, a single intravenous infusion of an equal amount of 0.9% saline before skin incision, followed by a continuous infusion at the same rate as the test group until 30 min before surgical cessation.
  Arms: Control group (placebo: saline)

SUMMARY:
This national, multi-center, randomized controlled study, through the study of intravenous injection of estaketamine in elderly patients undergoing surgery, is expected to explore whether estaketamine can improve the acute postoperative pain of elderly patients undergoing surgery and reduce the incidence of postoperative depression and delirium.

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged > 65 years old, no gender limitation;
* 2) patients undergoing elective thoracic, abdominal and orthopedic surgery;
* 3) ASA score is Class I-Class ~III;
* 4) 18 kg/ m2<BMI<30kg/m2；
* 5) The operation time is estimated to be 2 h-4 h;
* 6) Know clearly and voluntarily participate in this study, and sign informed consent form by oneself.

Exclusion Criteria:

* 1) patients with severe chronic pain;
* 2) Anemia or thrombocytopenia, Hb < 90 g/L, PLT < 80 × 109/L;
* 3) Severe liver dysfunction, AST and/or ALT≥2.5×ULN, and TBIL ≥ 1.5 × ULN;
* 4) severe renal dysfunction, blood creatinine is greater than the upper limit of normal;
* 5) Severe cardiovascular history (such as myocardial ischemia, heart failure and arrhythmia); Angina pectoris (unstable angina pectoris) caused by insufficient blood supply to the coronary vessels of the heart, or myocardial infarction in the past 6 months; QT interval prolongation (≥460ms in males and ≥ 470 ms in females);
* 6) Patients with hypertension whose blood pressure is not satisfactorily controlled by antihypertensive drugs (systolic blood pressure in sitting position during screening stage ≥180 mmHg, and/or diastolic blood pressure during screening stage ≥ 100 mmHg);
* 7) Patients with craniocerebral injury, possible intracranial hypertension, cerebral aneurysm, cerebrovascular accident history and central nervous system disease history;
* 8) patients with glaucoma or serious increase in intraocular pressure risk;
* 9) patients with mental system diseases (schizophrenia, mania, bipolar disorder, mental disorder, etc.) and drug history and cognitive dysfunction; History of cognitive psychiatric disorders such as postoperative delirium; Pregnant or lactating women;
* 10) high risk surgery, is expected to enter the ICU after surgery;
* 11) to moxa ketamine hydrochloride and its drug components allergy or taboo;
* 12) Being a subject and having participated in clinical trials for other drugs in the past three months;
* 13) There is communication disorder;
* 14) Patients considered by the investigator to be ineligible for participation in this trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
NRS pain score at the 24th hour after operation. | 24th hour after operation
  NRS pain score at the 24th hour after operation.

SECONDARY OUTCOMES:
NRS pain scores at the 2nd hour, 48th hour and 72nd hour after operation. | the 2nd hour, 48th hour and 72nd hour after operation.
  NRS pain scores at the 2nd hour, 48th hour and 72nd hour after operation.
The evaluation of APS-POQ-R questionnaire at 24 hours, 48 hours and 72 hours after operation. | 24 hours, 48 hours and 72 hours after operation.
  The evaluation of APS-POQ-R questionnaire at 24 hours, 48 hours and 72 hours after operation.
The consumption of anesthetic and analgesic drugs during and within 72 hours after operation. | during and within 72 hours after operation.
The scores of Montgomery Depression Scale at 24th hour, 48th hour and 72nd hour after operation. | 24th hour, 48th hour and 72nd hour after operation.
The score of GAD-7 anxiety scale 72 hours after operation. The incidence of delirium within 72 hours after operation | 72 hours after operation
The incidence of delirium within 72 hours after operation | 72 hours after operation
The incidence of adverse events during and within 72 hours after operation. | 72 hours after operation.